CLINICAL TRIAL: NCT03384680
Title: A Study on Symptom Collection of Patients With Lung Cancer.
Brief Title: Symptom Collection of Lung Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seong-Gyu Ko (Other)
Responsible Party: Sponsor-Investigator, Seong-Gyu Ko, Prof., Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Other Study IDs: KCRD_Lung cancer_Symptoms
Record Dates: First submitted 2017-12-20; First posted 2017-12-27 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is conducted to collect the symptoms of lung cancer patients and to observe the relationship with proteomics.

ELIGIBILITY:
Inclusion Criteria:

* Adult over 18 years old
* Patients are scheduled for surgery with lung cancer diagnosis.
* ECOG status score 0 to 2
* Individual who can read and understand Korean
* Participant is willing and able to give informed consent for participation in the study

Exclusion Criteria:

* Patient who was diagnosed with lung cancer in the past.
* Individuals who are judged inappropriate for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lung cancer who are scheduled for surgery will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-03-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Pattern identification | For 1 year
  Pattern identification by Body constitution questionnaire(BCQ) BCQ(+) is a questionnaire that is comprised of nineteen questions with one-to-five rating scales, making the range of total score to be between nineteen and ninety-five points with the cut-off score of 30.5 points for Yang-Xu.
  BCQ(-) is composed of another set of nineteen questions with the same five-point Likert scales, with the cut-off score of 29.5 points for Yin-Xu.
  BCQ(s) consists of twenty-three questions with the same Likert scale cut-off score of 26.5 points for Stasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cho W, Kim JH, Jeong M, Kim MS, Lee J, Son H, Cheon C, Park S, Ko SG. Pattern identification of lung cancer patients based on body constitution questionnaires (BCQ) and glycoproteomics for precision medicine. Medicine (Baltimore). 2019 Jun;98(24):e16035. doi: 10.1097/MD.0000000000016035. PMID 31192960